CLINICAL TRIAL: NCT00923416
Title: A Prospective Quantification of Patient-Reported Adverse Events Following Trans-Rectal Ultrasound-Guided Intra-Prostatic Marker Insertion
Brief Title: Trans-Rectal Ultrasound-Guided (TRUS) Adverse Events
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: UHN REB 08-0136-CE
Record Dates: First submitted 2009-06-16; First posted 2009-06-18 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Prostate Cancer
Keywords: Intra-Prostate Markers; Transrectal Ultrasound; Prostate Cancer Patients
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prostate Cancer

SUMMARY:
The goal of this study is to identify any side effects caused by the implanting of markers via the rectum. The investigators will also try to determine if any other factors (such as the position of the markers) influence the risk of side effects. The study procedures consist of two questionnaires:The first will be completed immediately after the marker implantation and the second questionnaire will be completed during your radiotherapy planning.

DETAILED DESCRIPTION:
Precise localisation of target organs has become increasingly important with the routine use of steep dose gradients from conformal and intensity modulated radiotherapy. This is particularly challenging when soft tissue target organs, such as the prostate, displace relative to bony anatomy. Although novel imaging techniques are being developed for the direct visualisation of such soft tissue structures, contrast and image quality is currently limited. However, the use of radio-opaque intra-prostatic fiducial markers(IPM) during high dose radiotherapy has proven very effective in terms of improving accuracy, and decreasing toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Have biopsy confirmed prostate cancer (any risk category)
* Have 3 intra-prostatic markers inserted at PMH prior to radiotherapy
* Be willing to provide written informed consent
* Be willing to complete the adverse event questionnaires

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate Cancer Patients who has trans-rectal ultrasound-guided implantation of intra-prostatic markers for radiotherapy treatment
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2008-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Quantify adverse events reported by prostate patients following trans-rectal ultrasound-guided implantation of intra-prostatic markers for RT | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tara Rosewall, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada